CLINICAL TRIAL: NCT00875797
Title: Comparison of Effect of Enteral Versus Parenteral Glutamine Supplement on Intestinal Permeability and Outcome of Critically Ill Patients
Brief Title: Enteral Versus Parenteral Glutamine Supplement
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Termination due to interim analysis results, inclusion problems in small ICUs.
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Lidija Kompan, MD, PhD, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P4-0092: onko
Record Dates: First submitted 2009-04-02; First posted 2009-04-03 (Estimated); Results first posted 2014-01-16 (Estimated); Last update posted 2014-01-16 (Estimated); Status verified 2013-12

CONDITIONS: Critically Ill
Keywords: enteral; parenteral; glutamine; intestinal permeability; infection
MeSH Terms: conditions — Critical Illness; Infections | interventions — alanylglutamine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- parentral glutamine (Active Comparator): parenteral glutamine given in central venous line in dose up to 30 g par day
  Interventions: Dietary Supplement: parenteral glutamine
- entral glutamine (Experimental): enteral glutamine given through gastric tube in a dose up to 30 g per day
  Interventions: Dietary Supplement: enteral glutamine

INTERVENTIONS:
Dietary Supplement: parenteral glutamine — Dipeptiven, Fresenius Kabi, Graz, Austria was given intravenously through central venous line in a dose up to 30 g per day
  Other Names: Dipeptiven, Fresenius Kabi, Graz, Austria
  Arms: parentral glutamine
Dietary Supplement: enteral glutamine — Alitraq, Abbott Laboratories, B.W. Zwolle, the Netherlands was given via nasogastric tube as continuous infusion of enteral diet, dose up to 30 g per day
  Other Names: Alitraq, Abbott Laboratories, B.W. Zwolle, the Netherlands
  Arms: entral glutamine

SUMMARY:
Glutamine is a major fuel for the intestinal tract and immune cells and therefore affects the intestinal permeability (IP) and infection rate at critically ill patients. The preferential route of glutamine supplementation at critically ill patients still remains open. Therefore the researchers will investigate IP, infection rate and treatment outcome at patients supplemented with either parenteral or enteral glutamine.

A prospective randomized single blind study is performed at mechanically ventilated. Patients were randomly assigned to either parenteral (group P) or enteral (group E) glutamine supplemented group. Early enteral feeding is started in both groups. Patients are/will be treated with glutamine for five days. IP will be measured using lactulose/mannitol test (L/M) on the fourth day.

DETAILED DESCRIPTION:
The patients who fulfilled the described criteria were randomly assigned to groups P or E using sequentially numbered containers for concealed randomization. Those in group P received the continuous infusion of parenteral glutamine dipeptide supplement (Dipeptiven 100ml, Fresenius Kabi) and were fed enterally with a standard commercial enteral polymeric diet without added glutamine (Ensure, Abbott Ross). The patients in group E received the enteral glutamine supplement as continuous administration of a standard commercial enteral diet supplemented with glutamine (Alitraq, Abbott Ross). The dose of the enteral glutamine, in a form of a free acid in this diet, depended on the volume of enteral food. Both groups of patients were treated with the glutamine supplement for five days. The other therapeutic procedures did not differ between the groups. All the patients were on continuous gastric feeding for 20 hours daily, starting with 20ml/hour. The enteral nutrition was started in 24 hours following admission. The gastric residual was measured three times daily, and when less than 250ml, the feeding volume was gradually increased up to 100ml/hour. If needed from day two onwards, the patients in all three groups received additional parenteral amino acid and glucose solutions to reach the goal 20kcal/kg/day and 0.15g nitrogen/kg/day.

Intestinal permeability (IP) was measured on day 4 using the lactulose/mannitol (L/M) test. For the study purpose, the patients were fasted 6 hours before the test. The test was performed with 5g of mannitol (M) and 10g of lactulose (L) mixed in 100ml of water. The mixture was given as a bolus via nasogastric tube. At the same time, 4ml of 20% chlorhexidine was added into an empty urine bag. The urine was collected in this bag for six hours. Then 5ml of urine was sampled from the bag and stored at -20˚C until analysis. Two hours after the test enteral feeding via nasogastric tube was started. Urinary L and M were determined simultaneously with thin-layer chromatography14, a new method in our laboratory for lactulose and mannitol determination. The method enabled determination of lactulose and mannitol in urine on the same amino HPTLC plate after densitometric quantification of lactulose by use of fluorescence mode, and mannitol by use of absorption mode after detection with AgNO3 reagent. The new method resulted in shorter analysis time, lower consumption of chemicals and HPTLC plates, increased sensitivity (lower limits of detection) and fewer problems with interfering compounds at determination of lactulose than the previously used two separate methods for determination of both analytes.14 The separation and quantification using this method are highly reproducible, yielding standard errors of less than 2.5% for retention times and less than 3.5% for quantitation.15,16 The investigators in the laboratory were blinded for the study groups. L/M index was calculated from urinary concentrations (c) of L and M using the following formula: L/M = c L / (c M x 2). L/M test was not performed at the beginning of the study because unstable trauma and septic patients were also included in the study, and at these patients, urine collection is difficult to perform.

Nosocomial infections were recorded during the entire ICU stay as recommended by the Centre for Disease Control in Atlanta.17,18 Nosocomial pneumonia was diagnosed when Hospital-Acquired Pneumonia Risk Index was 6 or more.19 The infections that were present upon admission or diagnosed within the first two days of ICU treatment were marked as acquired before ICU admission. All diagnosed infections were treated according to the results of microbiological tests and/or according to infection control guidelines. Acute inflammatory response was measured with C-reactive protein (CRP) levels. The blood samples for its determination were obtained at baseline and the end of the study.

Acute Physiology and Chronic Health Evaluation II (APACHE II) score was calculated upon admission. Each patient's ICU and hospital length of stay (LOS) and six month survival was recorded.

All participants were blinded to interventions. The ICU-staff was not blinded to group assignment, but they did not take part in the outcome assessment and on the other hand, the outcome assessors and laboratory personnel were blinded to group assignment.

ELIGIBILITY:
Inclusion Criteria:

* mechanically ventilated critically-ill patients
* older than 18 years
* staying in intensive care unit for at least 4 days

Exclusion Criteria:

* anuria
* intestinal insufficiency (obstruction, discontinuation of intestine or severe ileus)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2004-10; Primary Completion 2009-01 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jasna Uranjek, MD, Principal Investigator — General Hospital Slovenj Gradec
Locations (1):
- General Hospital Slovenj Gradec, Slovenj Gradec, Slovenia

REFERENCES:
- [Background] Luo M, Bazargan N, Griffith DP, Estivariz CF, Leader LM, Easley KA, Daignault NM, Hao L, Meddings JB, Galloway JR, Blumberg JB, Jones DP, Ziegler TR. Metabolic effects of enteral versus parenteral alanyl-glutamine dipeptide administration in critically ill patients receiving enteral feeding: a pilot study. Clin Nutr. 2008 Apr;27(2):297-306. doi: 10.1016/j.clnu.2007.12.003. Epub 2008 Feb 7. PMID 18258342

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Mechanically ventilated surgical and trauma critically-ill patients, older than 18 years, were enrolled in the study upon admission to ICU.
Pre-assignment Details: The patients with anuria or/and intestinal insufficiency (obstruction, discontinuation of intestine or severe paralytic ileus) were excluded from the study
Groups:
- Group P: Group P - group with parenterally supplemented glutamine
- Group E: Group E - group with enterally supplemented glutamine
Period: Overall Study
Arm/Group | Group P | Group E
Started | 45 | 45
Completed | 39 | 42
Not Completed | 6 | 3
Not completed — Protocol Violation | 6 | 3

BASELINE CHARACTERISTICS:
Population: mixed surgical ICU population
Groups:
- Parenteral Glutamine: parenteral glutamine supplementation
- Enteral Glutamine: enteral glutamine supplementation
- Total: Total of all reporting groups
Arm/Group | Parenteral Glutamine | Enteral Glutamine | Total
Number analyzed (Participants) | 45 | 45 | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1
  Between 18 and 65 years | 32 | 32 | 64
  >=65 years | 13 | 12 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.97 (12.90) | 51.40 (20.19) | 53.60 (17.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 14 | 29
  Male | 30 | 31 | 61

OUTCOME MEASURES:

1. Primary Outcome: Intestinal Permeability - Lactulose-mannitol(L/M)Test
Description: Measurement of intestinal permeability using lactulose-mannitol test (L/M test).
  Intestinal permeability to sugars is an accurate test for detecting intestinal damage. Intestinal permeability of the epithelium to very small sugar molecules such as lactulose/mannitol may give useful information regarding the overall condition of the digestive tract.
  Mannitol is absorbed transcellularly and lactulose has a paracellular route of absorption. Reduction in mannitol absorption shows reduced surface area and increased lactulose absorption indicates a leaky gut.
  Lactulose and mannitol are given orally and later determined from the collected urine with HPTLC (high performance thin layer chromatography). The L/M ratio, as a result of lactulose-mannitol tests, is then calculated regarding urine lactulose and mannitol concentrations.
  Thus, with the lactulose/mannitol test the intestinal permeability changes due to different reasons can be evaluated.
Time Frame: 4 days after admission to intensive care unit
Measure: Mean (Standard Deviation); unit: L/M ratio
Groups:
- Group P - Parenteral Glutamine: Group P - group with parenterally supplemented glutamine
- Group E - Enteral Glutamine: Group E - group with enterally supplemented glutamine
Arm/Group | Group P - Parenteral Glutamine | Group E - Enteral Glutamine
Number analyzed (Participants) | 39 | 42
L/M ratio | 0.492 (0.68) | 0.521 (0.86)
Statistical Analysis 1: Comparison: Group P - Parenteral Glutamine vs Group E - Enteral Glutamine; Test type: Non-Inferiority or Equivalence — t-test; p = 0.05, t-test, 2 sided — p<0.05

2. Secondary Outcome: Infection Rate at Participants in Both Groups
Description: Number of infections that occured at participants during study.
Time Frame: participants were followed for the duration of ICU stay (average 3 weeks)
Measure: Number; unit: number of infections
Groups:
- Group - Enteral Glutamine: Group E - group with enterally supplemented glutamine
Arm/Group | Group P - Parenteral Glutamine | Group - Enteral Glutamine
Number analyzed (Participants) | 39 | 42
number of infections | 15 | 12
Statistical Analysis 1: Comparison: Group P - Parenteral Glutamine vs Group - Enteral Glutamine; Test type: Non-Inferiority or Equivalence — χ2 test; p = 0.05, Chi-squared — p<0.05; 2 degrees of freedom; percentage of infection = 20, Standard Deviation 10

3. Secondary Outcome: 6-month Survival
Description: Six month follow up
Time Frame: 6 month
Measure: Number; unit: participants
Groups:
- Group P - Parenteral Glutamine: parenteral glutamine supplementation
- Group E - Enteral Glutamine: enteral glutamine supplementation
Arm/Group | Group P - Parenteral Glutamine | Group E - Enteral Glutamine
Number analyzed (Participants) | 39 | 42
participants | 31 | 36
Statistical Analysis 1: Comparison: Group P - Parenteral Glutamine vs Group E - Enteral Glutamine; Chi-square; Test type: Superiority or Other; p < 0.05, Chi-squared, Corrected — p<0.05; 2-degrees of freedom; percentage of survivers = 80

ADVERSE EVENTS:
Arm/Group | Group P | Group E
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/45
Other Adverse Events (participants affected / at risk) | 0/45 | 0/45

LIMITATIONS AND CAVEATS:
Termination due to small sample size for nutritional pilot study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No